CLINICAL TRIAL: NCT04438304
Title: Positron Emission Tomography Imaging of Participants With Known or Suspected Neuroendocrine Tumours Using 64Cu SARTATE: A Multi-Centre, Single Arm, Non-Randomised, Blinded-Review, Phase II Study
Brief Title: A Diagnostic Imaging Study of 64Cu-SARTATE Using PET on Patients With Known or Suspected Neuroendocrine Tumors (DISCO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLS07
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 64Cu-SARTATE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 64Cu-SARTATE will be administered at a fixed administration dose of 200 MBq (5.4 mCi) given as a single bolus intravenous injection.
  Interventions: Drug: 64Cu-SARTATE

INTERVENTIONS:
Drug: 64Cu-SARTATE — 64Cu-SARTATE will be administered at a fixed administration dose, single bolus intravenous injection, peptide mass not exceeding 60µg.
  Other Names: 64Cu-MeCOSar-Octreotate

SUMMARY:
The purpose of this study is to assess the performance of imaging agent 64Cu-SARTATE in participants with known or suspected Gastroenteropancreatic (GEP) Neuroendocrine Tumors (NETs) as a potential new way to help diagnose NETs.

DETAILED DESCRIPTION:
Up to 63 participants will be recruited in this study and who are confirmed or suspected to have NETs based on biochemical evidence or that of conventional anatomical or molecular imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Age at enrolment ≥ 18 years;
3. Life expectancy ≥ 12 weeks;
4. Known diagnosis of GEP NET or suspicion of GEP NET based on axial imaging (e.g. on CT and/or MRI and/or FDG) and/or biochemical evidence of NET;
5. Adequate recovery from acute toxic effects of any prior therapy;
6. Adequate renal function (eGFR >30 ml/min);
7. Pre-study 68Ga-DOTATATE PET/CT scan performed within 5 weeks, but not closer than 6 hours prior to the administration of 64Cu-SARTATE;

Exclusion Criteria:

1. Female participant who are pregnant or lactating;
2. Male or female participant of childbearing potential not willing to practice an effective method of birth control while participating on the study to avoid possible damage to the foetus. Abstinence is considered acceptable;
3. Participant has received any treatment (including experimental treatment) for their NET in the interval between 68Ga-DOTATATE PET/CT and 64Cu SARTATE PET/CT scan;
4. Any serious medical condition or extenuating circumstance which the investigator believes may interfere with the procedures or evaluations of the study;
5. History of other active malignancy within the last 2 years the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, in-situ carcinoma of the uterine cervix, or prostate cancer that is controlled by hormone therapy (patients may continue hormone therapy while on study).
6. Active oncologic therapy within 8 weeks prior to the 68GaDOTATATE PET/CT scan (long-acting somatostatin analogues are permitted and not considered active oncological treatment);
7. Participants with diffuse or infiltrative hepatic involvement based on the pre-study 68Ga-DOTATATE PET/CT scan;
8. Participants with extensive marrow/skeletal involvement (>20 lesions) based on the pre-study 68Ga-DOTATATE PET/CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Comparison of diagnostic performance of 64Cu-SARTATE to that of 68Ga-DOTATATE on a per-lesion basis for discordant findings | At 4 hours post administration of 64Cu-SARTATE
  Sensitivity and specificity on the 4-hour 64Cu-SARTATE PET/CT compared to 68Ga-DOTATATE PET/CT.
Comparison of diagnostic performance of 64Cu-SARTATE to that of 68Ga-DOTATATE on a per-lesion basis for discordant findings | At 20 hours post administration of 64Cu-SARTATE
  Sensitivity and Specificity on the 20-hour 64Cu-SARTATE PET/CT compared to 68Ga-DOTATATE PET/CT.
Comparison of diagnostic performance of 64Cu-SARTATE to that of 68Ga-DOTATATE on a per-lesion basis for discordant findings | At 4 and 20 hours post administration of 64Cu-SARTATE
  Lesion detection rate on composite of 4-hour and 20-hour 64Cu-SARTATE PET/CT compared to 68Ga-DOTATATE PET/CT.
To assess the proportion of concordance between 4-hour 64Cu-SARTATE to that of 68Ga-DOTATATE | At 4 hours post administration of 64Cu-SARTATE
  Concordance measured on a per-lesion basis

SECONDARY OUTCOMES:
To compare the diagnostic performance of 64Cu-SARTATE to 68Ga-DOTATATE on a per-participant basis in participants with suspected disease only. | At 4 hours and 20 hours post administration of 64Cu-SARTATE
  1. Sensitivity and specificity of the 4-hour 64Cu-SARTATE PET/CT compared to 68Ga-DOTATATE PET/CT.
  2. Sensitivity and specificity of the 20-hour 64Cu-SARTATE PET/CT compared to 68Ga-DOTATATE PET/CT.
Incidence of adverse events related to 64Cu-SARTATE | 1 week post administration of 64Cu-SARTATE
  Adverse events will be graded using the national cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria